CLINICAL TRIAL: NCT06434610
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of B013 Combined With Paclitaxel in the Treatment of Platinum-resistant Recurrent Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer.
Brief Title: A Study of B013 in Combination With Paclitaxel in Patients With Platinum-resistant Recurrent Ovarian Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH-B013-201
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B013 (Experimental)
  Interventions: Drug: B013; Drug: Paclitaxel
- Placebo (Placebo Comparator)
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: B013 — B013: The subjects will receive IV dose of B013 600 mg on Day 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Arms: B013
Drug: Paclitaxel — Paclitaxel: 80 mg/m^2 is administered weekly on Day 1, 8, 15 of each 28-day cycle.
Drug: Placebo — Placebo: The subjects will receive IV dose of placebo matched to B013 on Day 1 and 15 of the first 28-day cycle, then on Day 1 of each subsequent 28-day cycle.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of B013 in patients with platinum-resistant recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in this study and sign informed consent form;
2. Ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by histopathological examination and meeting the criteria for platinum resistance recurrence;
3. ECOG performance status of 0 or 1；
4. Expected survival > 12 weeks;
5. The subject has at least one measurable lesion;
6. Normal function of major organs;
7. The fertile subjects agree to use reliable contraception from signing the informed consent to at least 6 months after the last dose.

Exclusion Criteria:

1. Subjects who have received prescribed treatment previously;
2. Subjects who are still using anti-tumor traditional Chinese patent medicines at the time of signing informed consent;
3. Subjects with known central nervous system metastasis and multiple bone metastasis;
4. Subjects who had clinical symptoms of pleural effusion, pericardial effusion or ascites before randomization and needed puncture drainage, or had received puncture drainage within the previous 2 weeks;
5. Have a history of other malignant tumors within 5 years before signing the informed consent;
6. Subjects with prescribed cardiovascular diseases;
7. Subjects with infections requiring intravenous antibiotic infusion within 2 weeks prior to randomization;
8. Had severe lung disease before randomization;
9. Before randomization, the peripheral nerve toxicity of previous anti-tumor treatment was > grade 2, and other reversible toxicity was > grade 1;
10. Subjects who had undergone surgery within 28 days prior to randomization and did not recover from adverse effects of surgery;
11. Subjects who participated in clinical trials within 30 days prior to randomization and received other unmarketed investigational drugs;
12. Subjects who are known to be allergic to any component of B013 or paclitaxel.
13. Subjects with a known history of substance abuse, alcohol or drug use; Subjects with a known history of neurological or psychiatric disorders;
14. Female subjects who are pregnant or breastfeeding;
15. Other situations determined by the researchers and/or sponsors as unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 2 years
  From the date of randomization to the date of progression disease or death , whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Disease control rate (DCR) | Approximately 2 years
  DCR was defined as the percentage of participants who have achieved complete response, partial response and stable disease.
Duration of remission (DOR) | Approximately 5 years
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause.
Overall Survival (OS) | Approximately 2 years
  Determination of the overall survival times of all participants.
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 5 years
  The incidence of adverse event (regardless of its relationship to study drug) will be classified using MedDRA and the severity of each adverse event will be graded using NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - XiangYa Hospital CentralSouth University, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Guangxi Medical University Cancer Hospital, Nanning
  - Fudan University Shanghai Cancer center, Shanghai
  - The Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Shananxi Provincial Cancer Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Yibin city second people's Hospital, Yibin
  - Henan Cancer Hospital, Zhengzhou